CLINICAL TRIAL: NCT06485609
Title: A Prospective, Randomized, Open, Parallel-controlled, Superiority Clinical Study of Radical Right Hemicolectomy Versus Radical Right Hemicolectomy Combined with Indocyanine Green Fluorescence Imaging Lymphatic Tracer Dissection for the Treatment of Right Colon Cancer
Brief Title: Clinical Study of Radical Right Hemicolectomy Versus Radical Right Hemicolectomy Combined with Indocyanine Green Fluorescence Imaging Lymphatic Tracer Dissection for the Treatment of Right Colon Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, chief physician, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU-36
Record Dates: First submitted 2024-05-07; First posted 2024-07-03 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- radical right hemicolectomy (No Intervention)
- radical right hemicolectomy combined with indocyanine green fluorescence imaging lymphatic tracer di (Experimental)
  Interventions: Procedure: radical right hemicolectomy combined with indocyanine green fluorescence imaging lymphatic tracer dissection

INTERVENTIONS:
Procedure: radical right hemicolectomy combined with indocyanine green fluorescence imaging lymphatic tracer dissection — radical right hemicolectomy combined with indocyanine green fluorescence imaging lymphatic tracer dissection
  Arms: radical right hemicolectomy combined with indocyanine green fluorescence imaging lymphatic tracer di

SUMMARY:
The purpose of this study is to explore the clinical outcomes of indocyanine green fluorescence using in laparoscopic radical right hemicolectomy for right colon cancer（T1-T4a N+ M0）

ELIGIBILITY:
Inclusion Criteria:

* 1. Age between 18 and 75 years old 2. Confirmed adenocarcinoma cancer pathologically 3. Location of tumor: from the cecum to the right third of the transverse colon 4. CT showed right colon cancer: T1-T4a N+ M0 5. ASA scores I-III 6. ECOG (Eastern Cooperative Oncology Group) scale performance status of 0 or 1 7. Patient or family member, able to understand the study protocol and willing to participate in the study, providing written informed consent

Exclusion Criteria:

* 1. Simultaneous or heterochronic multiple primary colon cancer 2. Patients with intestinal obstruction, intestinal perforation, intestinal bleeding, etc. requiring emergency surgery 3. Unsuitable for laparoscopic surgery (e.g., extensive adhesions due to previous major abdominal surgery; unsuitable for pneumoperitoneum for various reasons, etc.) 4. Pregnant or lactating women 5. Have a history of serious mental illness 6. History of iodine allergy 7. History of other malignant diseases within the last five years 8. History of prior neoadjuvant chemotherapy or radiation therapy 9. History of unstable angina or myocardial infarction within the last 6 months 10. History of continuous systemic corticosteroid use within one month

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2024-08-10 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival rate | 3 years

SECONDARY OUTCOMES:
Number of lymph nodes cleared | Immediately after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No